CLINICAL TRIAL: NCT01852383
Title: An Open Treatment Trial of Duloxetine in Elderly Patients With Dysthymic Disorder
Brief Title: Duloxetine Treatment in Elderly With Dysthymia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6143R
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-02

CONDITIONS: Depression; Dysthymic Disorder
Keywords: Duloxetine; Antidepressant; Depression; Dysthymic Disorder; Side Effects; Elderly
MeSH Terms: conditions — Depression; Dysthymic Disorder | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duloxetine (Experimental): A minimum 1-week psychotropic medication washout, and a washout of 3 weeks for fluoxetine and monoamine oxidase inhibitors(MAOIs), was required. Duloxetine was prescribed at 20 mg daily for the first week, 30 mg daily for the second week, then 60 mg daily for another 4 weeks. Patients could subsequently be raised to 90 mg daily for another 2-4 weeks and then to a maximum dose of 120 mg daily.
  At all visits, the study psychiatrist had the option of adjusting the dose based on clinical response and side effects.
  Administration was as a single a.m. dose.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Patients were evaluated weekly for the first 6 weeks and every two weeks for the next 6 weeks. At 0, 1, 4, 8, and 12 weeks, the study psychiatrist completed the Cornell Dysthymia Rating Scale , Clinical Global Impression (CGI) scale, and side effect ratings using the Treatment Emergent Symptom Scale. The research rater completed a SCID-P at baseline and the 24-item HAM-D at each visit, and the patient completed the Beck Depression Inventory-II at each visit.
  Adverse events: All adverse events and serious adverse events were documented.
  The maximum duration of delay before active treatment (medication or psychotherapy) was 1 week.
  Dropout: Patients who had a CGI score of 6 or 7 for two weeks during the second half of the study were dropped by the investigator from the trial.
  Other Names: Cymbalta

SUMMARY:
Dysthymic disorder (DD) denotes chronic depression with fewer symptoms than major depressive disorder (MDD), and it affects ~ 2-4 % of adults with a similar prevalence in the elderly. In the elderly, dysthymic disorder (DD) has been shown to be associated with suffering and disability. The differences between young adult and elderly DD patients indicate that findings obtained in young adults with DD cannot be extrapolated to elderly DD patients who need to be studied separately. Data from epidemiologic studies support this view. In contrast to the data in young adult DD patients, there is a paucity of controlled data on the treatment of elderly DD patients. In our center, a double-masked, placebo-controlled study of 91 elderly DD patients did not find significant superiority for fluoxetine over placebo with response rates of 27.3% for fluoxetine and 19.6% for placebo in intent-to-treat analyses, and response rates of 37.5% for fluoxetine and 23.1% for placebo in completer analyses. Given the relative failure of selective serotonin reuptake inhibitor (SSRIs) to treat geriatric DD effectively, the investigators decided to evaluate the dual reuptake inhibitor, venlafaxine.

The investigators earlier completed an investigator-initiated, open-label 12-week venlafaxine (Effexor XR) trial. Of 23 elderly DD patients, 18 completed the trial. Fourteen (60.9%) were responders in intent-to-treat analyses with the last observation carried forward, and 77.8% were responders in completer analyses. Nearly half the sample (47.8%) met criteria for remission. In the intent-to-treat sample, increased severity of depression at baseline was associated with superior response and the presence of cardiovascular disease was associated with poorer response. These results with venlafaxine indicate that further treatment studies of dual serotonin-norepinephrine reuptake inhibitors like duloxetine are warranted in elderly patients with dysthymic disorder.

DETAILED DESCRIPTION:
HYPOTHESES:

1. Duloxetine will reduce depressive symptomatology over a period of 12 weeks in elderly DD patients.
2. Duloxetine-treated dysthymic patients will have significant improvement in measures of overall functioning.

This pilot trial enrolled 30 patients ≥ 60 years old with dysthymic disorder. Patients were recruited by clinician referral and by radio or newspaper advertisements that offered free evaluation by experienced clinicians for participation in clinical trials in the Adult and Late Life Depression Clinic at the New York State Psychiatric Institute. After a telephone screen to rule out exclusions for enrollment in the clinic, a psychiatrist conducted a detailed evaluation and completed the Cumulative Illness Rating Scale (CIRS)-Geriatric [CIRS-G]. Patients with a provisional clinical diagnosis of dysthymic disorder were interviewed by a research rater (social worker or nurse) with the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) Axis I disorders- Patient edition (SCID-P). Based on the psychiatrist's evaluation and the SCID-P interview, a consensus DSM-IV diagnosis was made at a staff conference.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dysthymic disorder (SCID and DSM-IV)
* Age 60 - 95
* Mini-Mental State Score ≥ 24
* 24-item Hamilton Rating Scale for Depression score 12-25
* Willing and capable of giving informed consent

Exclusion Criteria:

* Current major depressive episode (SCID and DSM-IV)
* Alcohol or substance dependence during the last year (SCID and DSM-IV)
* Bipolar disorder, schizophrenia and other psychotic disorders(SCID and DSM-IV)
* Clinical stroke, dementia, Huntington's disease, epilepsy or other major neurological disease
* Acute unstable medical conditions
* Active suicidal ideation or plan
* Non-response to duloxetine (minimum 90 mg/day for 6 weeks) during the past year
* A positive urine drug screen for substances of abuse or dependence
* Sensitivity with intolerability to duloxetine
* Use of other medications that may interact with duloxetine, including inhibitors of cytochrome P450 1A2 (CYP1A2) and cytochrome P450 2D6 (CYP2D6), e.g., quinolone antibiotics and type 1-C anti-arrhythmics. Several antidepressant medications, including most SSRIs, are inhibitors of CYP2D6 but these medications are not permitted during this antidepressant treatment trial.
* Patients with hypertension (BP >140/90 mm Hg on 2 consecutive measurements). For patients with treated hypertension and BP >140/90, written approval must be obtained from patient's internist allowing them to participate in this study.
* Known liver damage or disease

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2010-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Nobler MS, Devanand DP, Kim MK, Fitzsimons LM, Singer TM, Turret N, Sackeim HA, Roose SP. Fluoxetine treatment of dysthymia in the elderly. J Clin Psychiatry. 1996 Jun;57(6):254-6. PMID 8666563
- [Background] Devanand DP, Juszczak N, Nobler MS, Turret N, Fitzsimons L, Sackeim HA, Roose SP. An open treatment trial of venlafaxine for elderly patients with dysthymic disorder. J Geriatr Psychiatry Neurol. 2004 Dec;17(4):219-24. doi: 10.1177/0891988704269818. PMID 15533993
- [Background] Devanand DP, Nobler MS, Cheng J, Turret N, Pelton GH, Roose SP, Sackeim HA. Randomized, double-blind, placebo-controlled trial of fluoxetine treatment for elderly patients with dysthymic disorder. Am J Geriatr Psychiatry. 2005 Jan;13(1):59-68. doi: 10.1176/appi.ajgp.13.1.59. PMID 15653941
- [Background] Wise TN, Wiltse CG, Iosifescu DV, Sheridan M, Xu JY, Raskin J. The safety and tolerability of duloxetine in depressed elderly patients with and without medical comorbidity. Int J Clin Pract. 2007 Aug;61(8):1283-93. doi: 10.1111/j.1742-1241.2007.01476.x. Epub 2007 Jun 22. PMID 17590215

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: A minimum 1-week psychotropic medication washout, and a washout of 3 weeks for fluoxetine and monoamine oxidase inhibitors(MAOIs), was required. Duloxetine was prescribed at 20 mg daily for the first week, 30 mg daily for the second week, then 60 mg daily for another 4 weeks. Patients could subsequently be raised to 90 mg daily for another 2-4 weeks and then to a maximum dose of 120 mg daily.
  At all visits, the study psychiatrist had the option of adjusting the dose based on clinical response and side effects. Dose increments at these specified time-points will not occur if the patient meets criteria for remission or develops intolerable side effects that require reducing the dose or stopping the medication.
  Administration will be as a single a.m. dose.
Period: Overall Study
Arm/Group | Duloxetine
Started | 30
Completed | 19
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression (HAM-D, 24-item) From 0 Weeks to 12 Weeks.
Description: The research rater completed the 24-item Hamilton Rating Scale for Depression (HAM-D) and documented the scores on each visit. Hamilton Rating Scale for Depression scores range from 0-50 with low scores or decreasing scores representing decreased severity and better outcome, and higher scores or increasing scores representing more severe depressive symptoms and a worse outcome. The change score was calculated by subtracting the Week 12 score from the Week 0 score.
Time Frame: Screen (0) and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 30
units on a scale | 8 (6.1)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, ANCOVA — Change from Week 0 to Week 12, not adjusted for multiple comparisons. Alpha=0.05 threshold for statistical significance

2. Other Pre Specified Outcome: Change in the Treatment Emergent Symptom Scale (TESS) Total Score From Week 0 to Week 12.
Description: The Treatment Emergent Symptom Scale (TESS) documents the presence of common side effects. There are 26 items and the total score range is 0-26. Low scores or decrease in scores represent less side effects and high scores or increase in scores represent more side effects. The change in side effect severity scores was calculated by subtracting the Week 12 score from the Week 0 score.
Time Frame: 0 and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 30
units on a scale | 5.2 (3.3)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.1, Corrlation — Change from Week 0 to Week 12, not adjusted for multiple comparisons. Alpha=0.05 threshold for statistical significance

3. Secondary Outcome: Change in Cornell Dysthymia Rating Scale Scores From Week 0 to Week 12
Description: Cornell Dysthymia Rating Scale scores from range 0-64. Lower or decreasing scores represent decreased severity and a better outcome, while higher or increasing scores represent more severe depression and a worse outcome. The change score was calculated by subtracting the Week 12 score from the Week 0 score.
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine: A minimum 1-week psychotropic medication washout, and a washout of 3 weeks for fluoxetine and monoamine oxidase inhibitors(MAOIs), was required. Duloxetine was prescribed at 20 mg daily for the first week, 30 mg daily for the second week, then 60 mg daily for another 4 weeks. Patients could subsequently be raised to 90 mg daily for another 2-4 weeks and then to a maximum dose of 120 mg daily.
  At all visits, the study psychiatrist had the option of adjusting the dose based on clinical response and side effects.
  Administration was as a single a.m. dose.
  Duloxetine: Patients were evaluated weekly for the first 6 weeks and every two weeks for the next 6 weeks. At 0, 1, 4, 8, and 12 weeks, the study psychiatrist completed the Cornell Dysthymia Rating Scale, Clinical Global Impression (CGI) scale, and side effect ratings using the Treatment Emergent Symptom Scale.
Arm/Group | Duloxetine
Number analyzed (Participants) | 30
units on a scale | 28.8 (10.4)
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; p < 0.001, ANCOVA — Change from Week 0 to Week 12, not adjusted for multiple comparisons. Alpha=0.05 threshold for statistical significance

4. Other Pre Specified Outcome: Maximum Duloxetine Oral Dose
Description: Maximum duloxetine oral dose
Time Frame: Week 0, 1, 2, 4, 6, 8, 10, 12
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Duloxetine
Number analyzed (Participants) | 30
mg | 101 (38.4)
Statistical Analysis 1: Comparison: Duloxetine; Correlation of maximum duloxetine dose with change in Hamilton Depression Rating Scale scores from 0 Weeks to 12 Weeks; Test type: Superiority or Other; p < .001, Pearson correlation — Pearson correlation coefficient. Not adjusted for multiple comparisons. Alpha=0.05 for statistical significance threshold

ADVERSE EVENTS:
Time Frame: Assessments were completed once a week throughout the 12-week trial.
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=30)
Constipation and Anorgasmia (Gastrointestinal disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes